CLINICAL TRIAL: NCT02706119
Title: Subcutaneous Versus Intravenous Basal Insulin in Non-critical Hospitalized Diabetic Patients That Receive Total Parenteral Nutrition
Brief Title: Insulin in Total Parenteral Nutrition
Acronym: INSUPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FPS-INSUPAR-2015-01
Record Dates: First submitted 2016-02-16; First posted 2016-03-11 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
Keywords: total parenteral nutrition; glargine insulin; insulin
MeSH Terms: conditions — Diabetes Mellitus; Hyperphagia; Insulin Resistance | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glargine insulin (Experimental): Single dose glargine insulin (basal component) + regular insulin within total parenteral nutrition (TPN) reservoir (prandial component). 50% of the total calculated dose of insulin is administered subcutaneously as single dose subcutaneous glargine insulin; remaining 50% of the total calculated dose of insulin is administered as regular insulin in the TPN reservoir. Interventions used: Intravenous glargine insulin, and regular insulin added to TPN bag
  Interventions: Drug: Subcutaneous glargine insulin; Drug: Regular insulin added to TPN bag
- Regular insulin (Active Comparator): Regular insulin added to TPN bag (basal + prandial component). The calculated total dose of insulin is administered as regular insulin in the TPN reservoir. Interventions used: Regular insulin added to TPN bag
  Interventions: Drug: Regular insulin added to TPN bag

INTERVENTIONS:
Drug: Subcutaneous glargine insulin — Glargine insuline is an insulin analogue which has a prolonged duration of action. Insulin glargine is obtained by recombinant DNA technology in Escherichia coli.
  Other Names: ATC code A10AE0; Lantus®; Abasaglar®
  Arms: Glargine insulin
Drug: Regular insulin added to TPN bag — Regular insulin is human insulin produced in Saccharomyces cerevisiae by recombinant DNA technology.
  Other Names: ATC code A10AB01; Actrapid®

SUMMARY:
Analyze the level of metabolic control achieved with a routine of regular insulin in the parenteral nutrition (PN) reservoir in addition to subcutaneous glargine insulin, versus only regular insulin in the PN reservoir.

DETAILED DESCRIPTION:
A pattern of basal insulin (using subcutaneous insulin glargine and regulating the stock as prandial), plus regular subcutaneous insulin as rescue, applied to total parenteral nutrition (TPN) should be as effective (glycemic control, variability) and safe (hypoglycemia) as the usual (regular insulin inside the TPN reservoir and subcutaneous insulin as rescue) in patients with type 2 diabetes critics.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Previously diagnosed with diabetes mellitus.
* Hospitalized but without intensive cares.
* Have indication of total parenteral nutritional support (TPN, meaning the covering over 70% of the estimated daily requirements intravenously) for a minimum of 5 days.
* Signature of informed consent.

Exclusion Criteria:

* Diabetes mellitus type 1, diabetes secondary to total pancreatectomy.
* Patients with intensive cares.
* Patients who have been prescribed TPN in intensive cares unity more than 48 hours before admission to hospitalization.
* Intradialytic parenteral nutrition.
* Patients under 18 or pregnant women.
* Patients with renal insufficiency stage 3 B (glomerular filtration rate < 45 mL / min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Basal blood glucose value before starting TPN | Before starting total parenteral nutrition
  Basal glucose value before starting TPN (in mg/dL).
Periodical blood glucose | Every 6h during 15 days of treatment
  All blood glucose values (in mg/dL) every 6 hours during 15 days of TPN infusion.
Variation of average blood glucose compared with total dose of insulin | In days 1, 5 and 15 of treatment
  Variation of average glucose (in mg/dL) compared with total dose of insulin (in mL), in days 1, 5 and 15 of treatment.
Number of hypoglycaemia | During TPN treatment up to 15 days
  Number of symptomatic and asymptomatic hypoglycaemia with blood glucose below 70 mg/dL during TPN treatment up to 15 days.
Number of severe hypoglycaemia | During TPN treatment up to 15 days
  Number of symptomatic and asymptomatic hypoglycaemia with blood glucose below 40 mg/dL during TPN treatment up to 15 days.
Hypoglycemia blood glucose values | Through study completion, an average of 15 days.
  If the patient refers typical symptoms of hypoglycemia, a measure of blood glucose (in mg/mL) is immediately taken to check the level
Hypoglycemia symptoms | Through study completion, an average of 15 days.
  If blood glucose <70 mg / dL, it is recorded whether or not the patient has symptoms consistent with hypoglycemia and how the episode terminates

SECONDARY OUTCOMES:
Standard deviation of blood glucose | At day 15 of treatment
  Standard deviation of blood glucose (SD): Expressed in milligrams per deciliter (in mg/dL).
Blood glucose coefficient of variation (CV) | At day 15 of treatment
  Coefficient of variation (CV): Expressed as a percentage (%). The ratio of the standard deviation of the blood glucoses values (in mg/dL) and the average blood glucose (in mg/dL), multiplied by 100.

OTHER OUTCOMES:
Infections related with catheter used in parenteral nutrition | At day 15 of treatment
  Investigator asses the occurrence of infectious complications in parenteral nutrition catheter. For the evaluation of the infections, temperature is collected daily and patient will perform a blood test weekly. It will be suspected infectious complication for any sudden onset of fever (usually "peaks"), with no other apparent source of infection.
Hypertriglyceridemia | Every 6h during 15 days of treatment.
  A determination above this value will be considered a complication: Hypertriglyceridemia ≥500 mg/dL
Hypernatremia | Every 6h during 15 days of treatment.
  A determination above this value will be considered a complication: Hypernatremia >150 mEq/L
Hyponatremia | Every 6h during 15 days of treatment.
  A determination below this value will be considered a complication: Hyponatremia <135 mEq/L
Hypokalemia | Every 6h during 15 days of treatment.
  A determination below this value will be considered a complication: Hypokalemia <3 mEq/L
Hypomagnesemia | Every 6h during 15 days of treatment.
  A determination below this value will be considered a complication: Hypomagnesemia <1.2 mg/dL
Hypophosphatemia | Every 6h during 15 days of treatment.
  A determination below this value will be considered a complication: Hypophosphatemia <2 mg/dL
Hyperchloremia | Every 6h during 15 days of treatment.
  A determination above this value will be considered a complication: Hyperchloremia >120 mEq/L
Hypocalcemia corrected calcium | Every 6h during 15 days of treatment.
  A determination below this value will be considered a complication: Hypocalcemia corrected calcium <8 mg/dL
Alteration of liver function markers | At day 7 and 15 of treatment
  Alteration of liver function markers is defined as an elevation twice higher than normal limits, according to each laboratory, of two of some of the following parameters (when previously normal): GGT, GOT, GPT, FA or total bilirubin, at least 7 days after initiating TPN.
Adverse events | At day 15 of treatment
  All adverse events (AEs) are recorded in the case report data since the moment when the patient signs the informed consent. These events will be defined following the organ classification database of MedDRA system.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira Fuster, PhD, Principal Investigator — Hospital Regional de Malaga
Locations (32):
- Spain (32):
  - Hospital Arquitecto Marcide-Naval, Ferrol, A Coruña
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital Son Llátzer, Palma de Mallorca, Balearic Islands
  - Hospital General Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Universitario Bellvitge, Barcelona
  - Hospital de Sant Joan Despi Moisès Broggi (Consorci Sanitari Integral), Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Soria-Utrilla V, Sasso CV, Romero-Zerbo SY, Adarve-Castro A, Lopez-Urdiales R, Herranz-Antolin S, Garcia-Almeida JM, Garcia-Malpartida K, Ferrer-Gomez M, Moreno-Borreguero A, Luengo-Perez LM, Alvarez-Hernandez J, Aragon-Valera C, Ocon-Breton MJ, Garcia-Manzanares A, Breton-Lesmes I, Serrano-Aguayo P, Perez-Ferre N, Lopez-Gomez JJ, Olivares-Alcolea J, Moreno-Martinez M, Tejera-Perez C, Garcia-Arias S, Abad-Gonzalez AL, Alhambra-Exposito MR, Zugasti-Murillo A, Parra-Barona J, Torrejon-Jaramillo S, Abuin J, Fernandez-Garcia JC, Olveira G; Nutrition Area of the Spanish Society of Endocrinology and Nutrition (SEEN). Biomarkers of oxidation, inflammation and intestinal permeability in persons with diabetes mellitus with parenteral nutrition: A multicenter randomized trial. Clin Nutr. 2025 Jan;44:155-164. doi: 10.1016/j.clnu.2024.11.044. Epub 2024 Dec 3. PMID 39672082
- [Derived] Olveira G, Abuin J, Lopez R, Herranz S, Garcia-Almeida JM, Garcia-Malpartida K, Ferrer M, Cancer E, Luengo-Perez LM, Alvarez J, Aragon C, Ocon MJ, Garcia-Manzanares A, Breton I, Serrano-Aguayo P, Perez-Ferre N, Lopez-Gomez JJ, Olivares J, Arraiza C, Tejera C, Martin JD, Garcia S, Abad AL, Alhambra MR, Zugasti A, Parra J, Torrejon S, Tapia MJ. Regular insulin added to total parenteral nutrition vs subcutaneous glargine in non-critically ill diabetic inpatients, a multicenter randomized clinical trial: INSUPAR trial. Clin Nutr. 2020 Feb;39(2):388-394. doi: 10.1016/j.clnu.2019.02.036. Epub 2019 Mar 20. PMID 30930133